CLINICAL TRIAL: NCT01975948
Title: Evaluation of a Mental Health Physician Support Program in Nova Scotia: Impact on Patient Outcomes and Stigmatization
Brief Title: Evaluation of a Mental Health Physician Support Program in Nova Scotia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Bianca Horner, Primary Mental Healthcare Education Leader, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CDHA-RS/2014-150
Record Dates: First submitted 2013-10-21; First posted 2013-11-05 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Major Depressive Disorder
Keywords: Mental Health; Education and Practice Support Program; Depression; Primary Care; Skill-based training; Patient centered outcomes
MeSH Terms: conditions — Depressive Disorder, Major; Psychological Well-Being; Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Mental Health PSP: Physicians (Experimental): Physicians training in Adult Mental Health Practice Support Program
  Interventions: Other: Mental Health Practice Support Program
- Treatment as Usual: Physicians (Active Comparator): Those administering treatment as usual for depression
  Interventions: Other: Treatment as Usual
- Mental Health PSP: Patients (Experimental): Those belonging to a physician who has completed the Adult Mental Health Practice Support Program training.
  Interventions: Other: Mental Health Practice Support Program
- Treatment as Usual: Patients (Active Comparator): Those receiving treatment as usual for depression
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: Mental Health Practice Support Program — 1. training and (2) practice support.
     * Three half day workshop sessions over a 24 week period.
     * Practice support:
       3 evidence based Supported Self Management tools (Cognitive Behavioral Interpersonal Skills Manual,Bounceback program, Antidepressant Skills Workbook), and Practice support coordinator provides guidance to incorporate newly acquired tools, skills, and processes
  Arms: Mental Health PSP: Patients; Mental Health PSP: Physicians
Other: Treatment as Usual — Physicians manage patients with depression as usual
  Arms: Treatment as Usual: Patients; Treatment as Usual: Physicians

SUMMARY:
The aim of this study is to test the program's effectiveness in a primary care setting in reducing stigma among medical personnel, increasing the comfort level of physicians and staff in providing care to those living with mental illness, and in improving client well-being and mental health.

DETAILED DESCRIPTION:
Skill-based approaches are effective in reducing stigma in health professionals.

Overview: The Nova Scotia (NS) Department of Health and Wellness and the Mental Health Commission of Canada launched a demonstration project in NS-Adult Mental Health Practice Support Program. Originating in British Columbia (BC), it uses a novel learning platform which supports primary healthcare providers with treatment and management of mental illness. We hypothesized that enhanced skills in program participants would lead to increased comfort on the part of practitioners, diminished social distance and stigmatization; improved clinical outcomes and a reduction in healthcare costs.

This evaluation has three co-primary objectives:

* To determine whether the Mental Health Practice Support Program (PSP) leads to lower levels of stigma among physicians participating in the program.
* To determine whether participation in the Mental Health PSP leads to lower levels of stigma among medical office assistants (MOAs)
* To determine whether participation of physicians in the Mental Health PSP leads to greater improvement in depressive symptom ratings among patients they are treating for depression, compared to treatment as usual.

Two secondary objectives:

* To determine whether participation in the PSP leads to improved occupational functioning compared to treatment as usual.
* To assess the impact of participation in the Mental Health PSP on healthcare costs.

Four exploratory objectives:

* To assess physicians' confidence and comfort in the management of depression treatment
* To determine whether physician participation int he Mental Health PSP is associated with a reduced frequency of antidepressant prescribing.
* To determine whether the patients of physicians participating in the Mental Health PSP report higher levels of satisfaction with the treatment that they receive.
* To determine whether patients participation in the Mental Health PSP is associated with improved quality of life.

Methods: Seventy seven practices with one hundred and eleven community-based family physicians were recruited. Each practice was assigned a practice number. Each physician within the practice was assigned a unique identifier number. Individual practitioner or practice teams were randomly assigned to intervention or control groups. Randomization was stratified on the total number of physicians per practice, as well as urban or rural setting to ensure equal distribution of practice clusters and urban and rural groups. STATA, version 12 [College Station, TX, 2012] to generate the sequence for practice [cluster] randomization. Random numbers were generated from a binomial distribution with a probability of success of 0.5. Intervention group participants attended 3 half-day workshops with a "6- week action period" between workshops to practice learnings. Practice support was provided through diagnostic assessment tools, evidence based self-management tools, and on-site practice support coordinator support. A stigma-assessment tool, the Opening Minds Scale for Healthcare Providers (OMS-HC), was administered to both groups at intervention group pre-training, and post-training. Providers comfort and confidence in diagnosing and managing mental illness was also assessed, at comparable times.

Upon completion of the intervention group training, physicians from both groups were asked to identify 3 consecutive evaluable patients. Patients were enrolled and allocated to intervention or control groups as per their associated physician.

ELIGIBILITY:
Physician sample:

* A valid license to practice in Nova Scotia.
* The provision of informed consent.

Patient sample:

Inclusion Criteria:

* Depression defined by PHQ-9 score of > 10.
* > 18 years old.
* Able to read and speak English.
* Sufficiently intact cognitive functioning (physician judgement).
* Free of urgent or emergent medical or psychiatric issues e.g. unstable cardiovascular disease, suicidal ideation.

Exclusion Criteria:

* Not currently under treatment for depression either with an antidepressant medication or psychotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bianca A Lauria-Horner, MD, Principal Investigator — Associate Professor Dalhousie University Department of Psychiatry; Scott Patten, FRCP(C), PhD, Principal Investigator — Professor, Departments of Community Health Sciences and Psychiatry, Calgary, Alberta
Locations (1):
- Dalhousie University Department of Psychiatry, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Results will be distributed through publications in academic journals and presented at upcoming conferences, study sponsors and contributors: i.e. the Mental Health Commission of Canada, the Nova Scotia Department of Health and Wellness, Dalhousie University, the University of Calgary, Doctors of Nova Scotia, study participants, etc.
  Study Protocol, SAP, and Informed Consent will be shared. However when SAP is checked below in IPD sharing field, it will not allow to be saved (check-mark in SAP does not remain when save button is clicked).
  De-identified patient data will not be shared as we made a commitment to physicians that only the PI would have access to this information, even though de-identified, some were concerned that patients could still be identified.
Supporting Information: Study Protocol, ICF
Time Frame: Available as of August 21/2017 till December 31/2017
Access Criteria: Contact: Bianca Lauria-Horner hornerb@dal.ca

REFERENCES:
- [Derived] Lauria-Horner B, Beaulieu T, Knaak S, Weinerman R, Campbell H, Patten S. Controlled trial of the impact of a BC adult mental health practice support program (AMHPSP) on primary health care professionals' management of depression. BMC Fam Pract. 2018 Nov 28;19(1):183. doi: 10.1186/s12875-018-0862-y. PMID 30486799

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy seven practices with one hundred and eleven community-based family physicians were recruited between September 2013 and January 2014.
Pre-assignment Details: 285 participants were enrolled in the study: Physicians (n=111);Patients (n=129); Medical office Staff (MOAs) (n=45)
  MOA Group: MOAs excluded from outcome analysis due to inconsistent particpation and small sample size
Groups:
- Mental Health Practice Support Program;Physician Sample: Physician training in Adult Mental Health Practice Support Program
  Mental Health Practice Support Program: (1) training and (2) practice support.
  •Three half day workshop sessions over a 24 week period.
  •Practice support: 3 evidence based Supported Self Management tools (Cognitive Behavioral Interpersonal Skills Manual,Bounceback program, Antidepressant Skills Workbook), and Practice support coordinator provides guidance to incorporate newly acquired tools, skills, and processes
- Depression Treatment as Usual;Physician Sample: Treatment as Usual for Depression
  Depression Treatment as Usual: Physicians manage patients with depression as usual
- Mental Health Practice Support Program;Patient Sample: Patients were assigned to the same arm as their physician who were randomized to the Practice Support Program training. Patients were enrolled between June 2014-May 2015 with the last follow-up visit in November 2015
- Treatment as Usual: Patient Sample: Patients were assigned to the same arm as their physician, who were randomized to treating their patients as usual. Patients were enrolled between June 2014-May 2015 with the last follow-up visit in November 2015
Period: Overall Study
Arm/Group | Mental Health Practice Support Program;Physician Sample | Depression Treatment as Usual;Physician Sample | Mental Health Practice Support Program;Patient Sample | Treatment as Usual: Patient Sample
Started | 56 | 55 | 72 | 57
Completed | 39 | 34 | 65 | 51
Not Completed | 17 | 21 | 7 | 6
Not completed — Withdrawal by Subject | 17 | 21 | 7 | 6

BASELINE CHARACTERISTICS:
Population: It should be noted that baseline measures for the physician group are based on pre and post training completers (n=73). Patient data is based on those who completed at least one data time point (n=116).
Groups:
- Practice Support Program: Physician Sample: Physician training in Adult Mental Health Practice Support Program
  Mental Health Practice Support Program: (1) training and (2) practice support.
  •Three half day workshop sessions over a 24 week period.
  •Practice support: 3 evidence based Supported Self Management tools (Cognitive Behavioral Interpersonal Skills Manual,Bounceback program, Antidepressant Skills Workbook), and Practice support coordinator provides guidance to incorporate newly acquired tools, skills, and processes
- Treatment as Usual: Physician Sample: Treatment as Usual for Depression
  Depression Treatment as Usual: Physicians manage patients with depression as usual
- Practice Support Program: Patient Sample: Patients of physicians trained in the Adult Mental Health Practice Support Program.
  Inclusion criteria included >18 years of age, with a diagnosis of depression, PHQ-9 score of > 10, able to read and speak in English at grade 6 level, and intact cognitive functioning (physician judgment). Exclusion criteria included active treatment with antidepressants within 5 weeks and psychotherapy within 3 months of enrollment, and clinically judged urgent or emergent medical/psychiatric condition by their physician.
- Treatment as Usual: Patient Sample: Patients of physician who were randomized in the control group (TAU).
  Inclusion criteria included >18 years of age, with a diagnosis of depression, PHQ-9 score of > 10, able to read and speak in English at grade 6 level, and intact cognitive functioning (physician judgment). Exclusion criteria included active treatment with antidepressants within 5 weeks and psychotherapy within 3 months of enrollment, and clinically judged urgent or emergent medical/psychiatric condition by their physician.
- Total: Total of all reporting groups
Arm/Group | Practice Support Program: Physician Sample | Treatment as Usual: Physician Sample | Practice Support Program: Patient Sample | Treatment as Usual: Patient Sample | Total
Number analyzed (Participants) | 39 | 34 | 65 | 51 | 189
Age, Customized [Number; unit: participants] — Measures for the physician group are based on pre and post training completers (n=73).
  participants
    Physician 20-29years | 0 | 2 | NA — This section applies only to physician population | NA — This section applies only to physician population | NA — Total not calculated because data are not available (NA) in one or more arms.
    Physician 30-39years | 8 | 5 | NA — This section applies only to physician population | NA — This section applies only to physician population | NA — Total not calculated because data are not available (NA) in one or more arms.
    Physician 40-49years | 10 | 14 | NA — This section applies only to physician population | NA — This section applies only to physician population | NA — Total not calculated because data are not available (NA) in one or more arms.
    Physician 50-59years | 16 | 10 | NA — This section applies only to physician population | NA — This section applies only to physician population | NA — Total not calculated because data are not available (NA) in one or more arms.
    Physician 60-69years | 5 | 3 | NA — This section applies only to physician population | NA — This section applies only to physician population | NA — Total not calculated because data are not available (NA) in one or more arms.
Age, Customized [Count of Participants; unit: Participants] — Patient data is based on those who completed at least one data time point (n=116).
  Participants
    Patients 18-29 years | NA — This section applies only to patient population | NA — This section applies only to patient population | 11 | 12 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patients 30-39 years | NA — This section applies only to patient population | NA — This section applies only to patient population | 13 | 18 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patients 40-49 years | NA — This section applies only to patient population | NA — This section applies only to patient population | 14 | 8 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patients 50-59 years | NA — This section applies only to patient population | NA — This section applies only to patient population | 9 | 7 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patients 60-69 years | NA — This section applies only to patient population | NA — This section applies only to patient population | 9 | 3 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patients >70 years | NA — This section applies only to patient population | NA — This section applies only to patient population | 5 | 1 | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 45 | 40 | 127
  Male | 18 | 13 | 20 | 11 | 62
Region of Enrollment [Number; unit: participants]
  Canada | 39 | 34 | 65 | 51 | 189
Years in practice [Number; unit: participants] — Measures for the physician group are based on pre and post training completers (n=73).
  participants
    Less than 1 year | 0 | 2 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms.
    1-4years | 7 | 2 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms.
    5-9years | 3 | 3 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms.
    10-14years | 3 | 5 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms.
    15-19years | 1 | 6 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms.
    20-24years | 9 | 3 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms.
    25-29years | 9 | 7 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms.
    30 years or more | 5 | 6 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms.
Pattern of work [Number; unit: participants] — Measures for the physician group are based on pre and post training completers (n=73).
  participants
    Full time | 34 | 29 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms.
    Part time | 5 | 5 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms.
Practice type [Number; unit: participants] — Measures for the physician group are based on pre and post training completers (n=73)
  participants
    Solo practice | 9 | 5 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms
    2-physician practice | 8 | 5 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms
    Small gp practice (<5) | 16 | 8 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms
    Large gp practice (5+) | 5 | 16 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms
Unique patients/yr [Number; unit: participants] — Measures for the physician group are based on pre and post training completers (n=73)
  participants
    Fewer than 1,000 | 6 | 7 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms
    1,000-1,999 | 12 | 12 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms
    2,000-2,999 | 2 | 7 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms
    3,000 or more | 11 | 6 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms
    Other (hospitalist, locum, etc) | 2 | 0 | NA — This section applies only to physician group | NA — This section applies only to physician group | NA — Total not calculated because data are not available (NA) in one or more arms
Marital Status [Count of Participants; unit: Participants] — Patient data is based on those who completed at least one data time point (n=116).
  Participants
    Patients: Married/common-law | NA — This section applies only to patient population | NA — This section applies only to patient population | 33 | 32 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patients: Separated/divorced | NA — This section applies only to patient population | NA — This section applies only to patient population | 11 | 5 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patients: Never married | NA — This section applies only to patient population | NA — This section applies only to patient population | 17 | 10 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patients: Widowed | NA — This section applies only to patient population | NA — This section applies only to patient population | 0 | 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
Employment status [Count of Participants; unit: Participants] — Patient data is based on those who completed at least one data time point (n=116).
  Participants
    Patients: Employed full time | NA — This section applies only to patient population | NA — This section applies only to patient population | 27 | 26 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patients:Employed part time | NA — This section applies only to patient population | NA — This section applies only to patient population | 8 | 13 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patients:Unemployed but available to work | NA — This section applies only to patient population | NA — This section applies only to patient population | 5 | 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patients:Unemployed due to illness | NA — This section applies only to patient population | NA — This section applies only to patient population | 6 | 3 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patients:Retired/student/at-home/other | NA — This section applies only to patient population | NA — This section applies only to patient population | 5 | 15 | NA — Total not calculated because data are not available (NA) in one or more arms.
Education [Count of Participants; unit: Participants] — Patient data is based on those who completed at least one data time point (n=116).
  Participants
    Some elementary or high school | NA — This section applies only to patient population | NA — This section applies only to patient population | 8 | 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
    High school diploma | NA — This section applies only to patient population | NA — This section applies only to patient population | 14 | 6 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Some post-secondary | NA — This section applies only to patient population | NA — This section applies only to patient population | 5 | 10 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Post-secondary certificate/diploma | NA — This section applies only to patient population | NA — This section applies only to patient population | 14 | 17 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Post-secondary degree | NA — This section applies only to patient population | NA — This section applies only to patient population | 15 | 13 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Master's degree or higher | NA — This section applies only to patient population | NA — This section applies only to patient population | 5 | 1 | NA — Total not calculated because data are not available (NA) in one or more arms.
Mother tongue [Count of Participants; unit: Participants] — Patient data is based on those who completed at least one data time point (n=116).
  Participants
    Patient: English | NA — This section applies only to patient population | NA — This section applies only to patient population | 56 | 48 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patient: French | NA — This section applies only to patient population | NA — This section applies only to patient population | 3 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patient: Other | NA — This section applies only to patient population | NA — This section applies only to patient population | 2 | 1 | NA — Total not calculated because data are not available (NA) in one or more arms.
Who do you usually live with? [Count of Participants; unit: Participants] — Patient data is based on those who completed at least one data time point (n=116).
  Participants
    Patient: Husband/wife/steady partner | NA — This section applies only to patient population | NA — This section applies only to patient population | 18 | 17 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patient:Spouse partner and children | NA — This section applies only to patient population | NA — This section applies only to patient population | 15 | 19 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patient:Children (but no spouse/partner) | NA — This section applies only to patient population | NA — This section applies only to patient population | 4 | 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patient:Parents | NA — This section applies only to patient population | NA — This section applies only to patient population | 4 | 4 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patient:Alone | NA — This section applies only to patient population | NA — This section applies only to patient population | 13 | 6 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patient:Other | NA — This section applies only to patient population | NA — This section applies only to patient population | 6 | 1 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Depression Severity (Change in Patient Health Questionnaire-9 (PHQ-9) Score From Baseline
Description: The Patient Health Questionnaire-9 (PHQ-9) covers nine symptom-based Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for major depressive disorder. Scores range from 0-27, with higher scores indicating more severe depression severity. We compared between-group mean differences of PHQ-9 scores during follow-up, assessed as a group-by-time interaction. We used a multi-level mixed model analysis: physicians clustered within practices, patients clustered within their corresponding physicians, and longitudinal PHQ-9 ratings clustered within patients. The four follow-up time points were represented by indicator variables. The effect of the intervention was measured as an intervention by time interaction, and the time-by-group interaction was assessed using a likelihood ratio test.
Time Frame: Baseline, 1, 2, 3, and 6 months
Population: All participants with at least one follow-up data (n=116) were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mental Health PSP: Patients | Treatment as Usual: Patients
Number analyzed (Participants) | 65 | 51
units on a scale
  baseline | 16.43 (4.77) | 17.28 (4.12)
  1 month | 11.25 (5.82) | 10.39 (6.49)
  2 months | 9.72 (6.28) | 8.46 (6.47)
  3 months | 8.44 (6.15) | 7.55 (6.13)
  6 month | 6.78 (5.41) | 8.42 (6.57)
Statistical Analysis 1: Comparison: Mental Health PSP: Patients vs Treatment as Usual: Patients; One hundred evaluable patients per arm were needed to achieve 80% power to detect a PHQ-9 between-group difference in mean change of 2 points, significance level (α) .05, a two-sided test, and a standard deviation of 5 points. An intra cluster correlation of 0.05 for patient outcomes was used (Murphey et al), and an average cluster size: 3 patients/practice resulted in compensatory increase to 110 patients per arm. Under the assumption that attrition would be 33 % we needed 166 patients per arm; Test type: Other; p = .047, Mixed Models Analysis — Adjusted for baseline depressive symptoms and unemployment as covariates (p=.016), and non-completers (missing one or more points of follow up data)

2. Primary Outcome: Between Group Changes in Total Score on the Opening Minds Scale for Health Care Providers (OMS-HC)
Description: The Opening Minds Scale for Health Care Providers (OMS-HC) is a 15 item validated scale that also captures three main dimensions of stigma; negative attitudes, health professionals' own willingness to disclose/seek help for a mental illness, and preference for greater social distance. Items are rated on a 5-point scale: from strongly agree to strongly disagree. Total scores can range from 15 to 75 for the overall total score, 6 to 30, 4-29, 5-25 for sub-scales respectively. Total scores are averaged to result in mean scores range from 1 to 5 with lower scores indicating less stigma. This scale has been widely validated and used in evaluations of anti-stigma interventions in Canada. The analysis was conducted using a multi-level mixed model in which physicians were clustered within practices and stigma ratings were clustered within physicians (one or two observations per physician). The effect of the intervention was measured in this analysis as an intervention by time interaction.
Time Frame: Baseline and at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mental Health PSP: Physicians: Physician training in Adult Mental Health Practice Support Program
  Mental Health Practice Support Program: (1) training and (2) practice support.
  •Three half day workshop sessions over a 24 week period.
  •Practice support: 3 evidence based Supported Self Management tools (Cognitive Behavioral Interpersonal Skills Manual,Bounceback program, Antidepressant Skills Workbook), and Practice support coordinator provides guidance to incorporate newly acquired tools, skills, and processes
- Treatment as Usual: Physicians: Depression Treatment as Usual: Physicians manage patients with depression as usual
Arm/Group | Mental Health PSP: Physicians | Treatment as Usual: Physicians
Number analyzed (Participants) | 39 | 34
units on a scale
  OMS-HC Total Score Baseline | 2.21 (.40) | 2.11 (.35)
  OMS-HC Total Score 6 months | 2.07 (.46) | 2.07 (.38)
  Attitudes subscale:Baseline | 2.13 (.48) | 2.02 (.48)
  Attitudes subscale: 6 months | 1.97 (.49) | 1.9 (.51)
  Disclosure/help-seeking: Baselinr | 2.65 (.66) | 2.65 (.61)
  Disclosure/help-seeking: 6 months | 2.57 (.75) | 2.63 (.52)
  Social distance: Baseline | 1.95 (.46) | 1.77 (.39)
  Social distance : 6 months | 1.79 (.55) | 1.82 (.48)
Statistical Analysis 1: Comparison: Mental Health PSP: Physicians vs Treatment as Usual: Physicians; Our calculations indicated that 50 physicians in each of the two groups will provide >80% power to detect clinically significant reductions in stigma as assessed by OMS-HC change scores. Clinically meaningful was defined as a change of 3 points, derived on the basis of this being slightly better than what is usually seen in brief interventions; Test type: Other; p = 0.15, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mental Health PSP: Physicians vs Treatment as Usual: Physicians; Between Group Changes in subscale of the Opening Minds Scale for Health Care Providers (OMS-HC) measures three different dimensions of stigma: attitudes towards people with a mental illness (6 items); health care professionals' attitudes about disclosure of a mental illness/willingness to seek help for a mental illness (4 items), and preference for social distance (5 items). Items are rated on a 5-point scale. Mean scores can range from one to five with lower scores indicating less stigma; Test type: Other; p = .03, Mixed Models Analysis — OMS-HC analysis adjusted for practice size: P value applies to between group physicians reduction in one stigma domaine: preference for social distance; Cohen'd = .45

3. Secondary Outcome: Between Group Changes in Occupational Functioning From Baseline to 6 Months
Description: Lam's Employment Absence and Productivity Scale (LEAPS) is a 7 item scale that assesses workplace impact of major depression. Each item is rated on a 5-point Likert scale with the following response format: none of the time (0%), some of the time (25%), half the time (50%), most of the time (75%), or all the time (100%), scored as 0-4, respectively. Total scores can range from 0-28 with lower scores indicating less disruption.We compared between-group mean differences of LEAPs scores during follow-up, assessed as a group-by-time interaction. We used a multi-level mixed model analysis: physicians clustered within practices, patients clustered within their corresponding physicians, and longitudinal LEAPs ratings clustered within patients. The four follow-up time points were represented by indicator variables. The effect of the intervention was measured as an intervention by time interaction, and the time-by-group interaction was assessed using a likelihood ratio test.
Time Frame: Baseline, 1, 2, 3, and 6 months
Population: All participants with at least one follow-up data (n=116) were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mental Health PSP: Patients | Treatment as Usual: Patients
Number analyzed (Participants) | 65 | 51
units on a scale
  Baseline | 11.26 (5.80) | 12.76 (6.52)
  1 month | 7.67 (5.36) | 7.13 (5.96)
  2 months | 7.45 (6.21) | 7.16 (6.88)
  3 months | 5.54 (4.37) | 5.96 (5.06)
  6 months | 6.04 (5.79) | 6.03 (6.12)
Statistical Analysis 1: Comparison: Mental Health PSP: Patients vs Treatment as Usual: Patients; Test type: Other; p = .993, Mixed Models Analysis

4. Other Pre Specified Outcome: Between Group Change at 6 Months From Baseline in Physician Confidence and Comfort in Managing Mental Illness
Description: A modified version of a British Columbia (BC) developed survey, "Practice Support Program Pre-Post Learning Module Questionnaire" was used. Physician confidence was measured on a three point scale ranging from 'very confident' to 'not at all confident.' Mean scores were averaged and can range from one to three, with lower scores indicating higher confidence. Physicians were asked to their level of confidence to:
  * diagnose depression
  * screen for addictions
  * screen for other mental health conditions
  * treat depression
  * treat other mental health disorders
  * prescribe medications for mental health conditions
  * assess patients' problems and strengths
  * overall confidence in quality of mental health care provided
  * knowledge/awareness of non-pharmaceutical interventions
  * knowledge/awareness of regional mental health resources for patients
  Cronbach's alpha .84 at pre-test and .87 at post-test
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Practice Support Program: Physician Sample | Treatment as Usual: Physician Sample
Number analyzed (Participants) | 39 | 34
units on a scale
  Baseline Management of mental illness | 2.18 (.39) | 2.03 (.37)
  6 monthsManagement of mental illness | 1.80 (.36) | 2.12 (.40)
Statistical Analysis 1: Comparison: Practice Support Program: Physician Sample vs Treatment as Usual: Physician Sample; Test type: Other; p < .001, Mixed Models Analysis; Cohen'd = 1.48
Statistical Analysis 2: Comparison: Practice Support Program: Physician Sample vs Treatment as Usual: Physician Sample; Correlation between increases in Physician Comfort and Confidence in managing mental illness and Stigma Score; Test type: Other; p = .03, Generalized estimating equations (GEE); We used the slope of a regression line fit using generalized estimating equations (GEE) with an exchangeable correlation structure

5. Other Pre Specified Outcome: Between Group Change in Physician Confidence and Comfort With Non-program Specific Tools and Skills
Description: A modified version of a British Columbia (BC) developed survey "Practice Support Program Pre-Post Learning Module Questionnaire" was used. Physicians were also asked to rate their level of familiarity, confidence and comfort with a variety of non-program specific mental health tools and skills for assisting patients with mental health concerns (e.g., PHQ9 & PHQ2, AUDIT, SMME, MOCA, GAF, GAD-7). Physician confidence was measured on a three point scale ranging from 'very confident' to 'not at all confident. Mean scores were averaged and can range from one to three, with lower mean scores indicating higher levels of comfort, confidence and familiarity. Cronbach's alpha for physicia was .90 at pre-test and .91 at post-test,
  3
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mental Health PSP: Physicians | Treatment as Usual: Physicians
Number analyzed (Participants) | 39 | 34
units on a scale
  Baseline non-program specific mental health tools | 2.34 (.4) | 2.27 (.5)
  6 months non-program specific mental health tools | 1.81 (.4) | 2.32 (.48)
Statistical Analysis 1: Comparison: Mental Health PSP: Physicians vs Treatment as Usual: Physicians; Test type: Other; p < .001, Mixed Models Analysis; Cohen'd = 1.44
Statistical Analysis 2: Comparison: Mental Health PSP: Physicians vs Treatment as Usual: Physicians; Correlation between increases in Physician Comfort and Confidence with non-program specific tools and Stigma Score; Test type: Superiority; p = .476, Generalized estimating equations (GEE) — We used the slope of a regression line fit using generalized estimating equations (GEE) with an exchangeable correlation structure

6. Other Pre Specified Outcome: Between Group Change in Physician Confidence and Comfort With Program Specific Tools and Skills
Description: A modified version of a British Columbia (BC) developed survey, Practice Support Program Pre-Post Learning Module Questionnaire was used. Physicians were also asked to rate their level of familiarity, confidence and comfort with a variety of non-program specific mental health tools and skills for assisting patients with mental health concerns (e.g., CBIS manual, electronic hyperlinked mental health algorithm, Bounce Back program DVD, referrals for Bounce Back telephone coaching, ASW and coaching skills, Diagnostic Assessment Interview, Problem List Action Plan, CBIS resource list, CBIS skills handout, Family Physician Guide, and medication algorithm). Physician confidence was measured on a three point scale ranging from 'very confident' to 'not at all confident. Mean scores were averaged and can range from one to three, with lower mean scores indicating higher levels of comfort, confidence and familiarity. Cronbach's alpha was .98 at pre-test and .98 at post-test
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mental Health PSP: Physicians | Treatment as Usual: Physicians
Number analyzed (Participants) | 39 | 34
units on a scale
  Baseline program specific mental health tools | 2.82 (.31) | 2.80 (.20)
  6 months program specific mental health tools | 1.79 (.44) | 2.64 (.21)
Statistical Analysis 1: Comparison: Mental Health PSP: Physicians vs Treatment as Usual: Physicians; Test type: Superiority; p < .001, Mixed Models Analysis; Cohen'd = 3.25
Statistical Analysis 2: Comparison: Mental Health PSP: Physicians vs Treatment as Usual: Physicians; Correlation between increases in Physician Comfort and Confidence with program specific tools and Stigma Score; Test type: Superiority; p = .945, Generalized estimating equations (GEE) — We used the Spearman's correlation coefficient using the slope of a regression line fit using generalized estimating equations (GEE) with an exchangeable correlation structure

7. Other Pre Specified Outcome: Between Goup Change in Client Satisfaction Inventory (CSI) From Baseline to 6 Months
Description: The CSI is a 25-item scale to measure the degree or magnitude of client satisfaction with care received. Responses range from 1 to 7. Total raw scores range from 0 to 175, with higher scores representing higher levels of satisfaction. Total scores were averaged reducing the overall score to a 7-point scale. We compared between-group mean differences of CSI scores during follow-up, assessed as a group-by-time interaction. We used a multi-level mixed model analysis: physicians clustered within practices, patients clustered within their corresponding physicians, and longitudinal CSI ratings clustered within patients. The four follow-up time points were represented by indicator variables. The effect of the intervention was measured as an intervention by time interaction, and the time-by-group interaction was assessed using a likelihood ratio test.
Time Frame: Baseline, 1, 2,3, and 6 months
Population: All participants with at least one follow-up data (n=116) were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mental Health PSP: Patients | Treatment as Usual: Patients
Number analyzed (Participants) | 65 | 51
units on a scale
  Baseline | 6.3 (.51) | 6.1 (.87)
  I month | 6.1 (.79) | 6.1 (.95)
  2 months | 6.2 (.76) | 6.2 (.95)
  3 months | 6.1 (.93) | 6.1 (.91)
  6 months | 6.1 (.79) | 6.0 (1.0)
Statistical Analysis 1: Comparison: Mental Health PSP: Patients vs Treatment as Usual: Patients; Test type: Other; p = .742, Mixed Models Analysis

8. Other Pre Specified Outcome: Between Groups Changes in Quality of Life From Baseline to 6 Months.
Description: The Medical Outcomes Short Form (SF-36) assesses quality of life. All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible. Aggregate scores are compiled as a percentage of the total points possible, using the RAND scoring table.We ompared between-group mean differences of SF-36 scores during follow-up, assessed as a group-by-time interaction. We used a multi-level mixed model analysis: physicians clustered within practices, patients clustered within their corresponding physicians, and longitudinal SF-36 ratings clustered within patients. The four follow-up time points were represented by indicator variables. The effect of the intervention was measured as an intervention by time interaction, and the time-by-group interaction was assessed using a likelihood ratio test.
Time Frame: Baseline, 1, 2, 3 and 6 months
Population: All participants with at least one follow-up data (n=116) were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mental Health PSP: Patients | Treatment as Usual: Patients
Number analyzed (Participants) | 65 | 51
units on a scale
  Baseline | 54.03 (14.07) | 54.10 (12.92)
  1 month | 57.73 (17.09) | 62.33 (15.30)
  2 months | 61.77 (18.38) | 67.62 (15.59)
  3 months | 62.45 (21.76) | 66.99 (18.83)
  6 months | 67.09 (20.88) | 69.03 (21.26)
Statistical Analysis 1: Comparison: Mental Health PSP: Patients vs Treatment as Usual: Patients; Test type: Other; p = .543, Mixed Models Analysis

9. Other Pre Specified Outcome: Number of Patients That Were Prescribed Antidepressant (AD) at 6 Months
Description: We compared between group use of antidepressant in both groups using the Client Service Receipt Inventory questionnaire at 6 months.
Time Frame: 6 months
Population: All participants with at least one follow-up data (n=116) were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Mental Health PSP: Patients | Treatment as Usual: Patients
Number analyzed (Participants) | 65 | 51
Participants | 31 | 35
Statistical Analysis 1: Comparison: Mental Health PSP: Patients vs Treatment as Usual: Patients; Test type: Other; p = .009, Mixed Models Analysis

10. Other Pre Specified Outcome: Between Group Change in Sheehan Disability Scale (SDS)
Description: The SDS is a visual analog scale which asks respondents to rate from 0-10 the extent to which symptoms have disputed: a: work/school work; b) social life/leisure activities; c) family life/home responsibilities. Total scores can range from 0-30, with lower scores indicating less disruption. We ompared between-group mean differences of SDS scores during follow-up, assessed as a group-by-time interaction. We used a multi-level mixed model analysis: physicians clustered within practices, patients clustered within their corresponding physicians, and longitudinal SDS ratings clustered within patients. The four follow-up time points were represented by indicator variables. The effect of the intervention was measured as an intervention by time interaction, and the time-by-group interaction was assessed using a likelihood ratio test.
Time Frame: Baseline, 1, 2, 3, and 6 months
Population: All participants with at least one follow-up data (n=116) were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mental Health PSP: Patients | Treatment as Usual: Patients
Number analyzed (Participants) | 65 | 51
units on a scale
  Baseline | 18.87 (7.06) | 19.83 (6.20)
  1 month | 13.87 (8.19) | 13.03 (8.99)
  2 months | 13.74 (9.12) | 9.43 (8.95)
  3 months | 10.42 (9.34) | 8.28 (7.29)
  6 months | 7.64 (7.27) | 7.86 (8.46)
Statistical Analysis 1: Comparison: Mental Health PSP: Patients vs Treatment as Usual: Patients; Test type: Other; p = .213, Mixed Models Analysis

ADVERSE EVENTS:
Description: Serious and other adverse events were not monitored/assessed. The clinical skills and knowledge addressed in the training are standard approaches, involving cognitive and behavioral strategies. There are no risks associated with the implementation of these strategies.
Arm/Group | Mental Health PSP: Patients | Treatment as Usual: Patients
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Challenges in physician sample: 75% completed pre-post OMS-HC scale Physicians experienced challenges identifying study patients leading to small number of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No